CLINICAL TRIAL: NCT01166113
Title: A Phase I/II, Multi-center, Open Label Study of Pomalidomide, Cyclophosphamide and Prednisone (PCP) in Patients With Multiple Myeloma Relapsed and/or Refractory to Lenalidomide
Brief Title: Pomalidomide, Cyclophosphamide and Prednisone (PCP) in Patients With Multiple Myeloma (MM) Relapsed and/or Refractory to Lenalidomide
Acronym: PCP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PO0023; 2009-014850-13 (EudraCT Number)
Record Dates: First submitted 2010-07-16; First posted 2010-07-20 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma
Keywords: Pomalidomide; Relapsed/Refractory to Lenalidomide
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — pomalidomide; Cyclophosphamide; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PCP (Experimental)
  Interventions: Drug: Pomalidomide, Cyclophosphamide, Prednisone

INTERVENTIONS:
Drug: Pomalidomide, Cyclophosphamide, Prednisone — Induction
  This multicenter phase I followed by a phase II trial will evaluate the safety and efficacy of the combination Pomalidomide-Cyclophosphamide-Prednisone (PCP) in patients (pts) with MM relapsed/refractory to lenalidomide.
  In the phase I we assess the maximum tolerated dose (MTD) of PCP in 25% of pts. The first 4 pts are given the second dose level, accrual continues with 4 pts per dose level for a maximum of 24 pts.
  The dose level associated with an updated DLT is recommended for the next patient cohort.
  Each patient is assigned to a salvage therapy including Cyclophosphamide and Prednisone (both 50 mg every other d), and Pomalidomide at one of the following doses:1 mg/d;1.5 mg/d;2 mg/d;2.5 mg/d
  In the phase II a total of 43 pts will be treated with the MTD of PCP. Pts enrolled at the MTD during the phase I will be included in the Phase II trial.
  Maintenance (each cycle repeated every 28 d, until PD) Pomalidomide: 2.5 mg/d; Prednisone: 25 mg every other d

SUMMARY:
This study will evaluate if the combination of Pomalidomide, Cyclophosphamide and Prednisone is safe and provides benefits in patients with multiple myeloma relapsed and/or refractory to lenalidomide.

DETAILED DESCRIPTION:
This is a prospective multicenter phase I followed by a phase II trial designed to evaluate the safety and efficacy of the combination of Pomalidomide with Cyclophosphamide and Prednisone in patients with multiple myeloma relapsed and/or refractory to lenalidomide.

Patients will be evaluated at scheduled visits in up to 3 study periods: pre-treatment, treatment and long-term follow-up (LTFU).

The pre-treatment period includes: screening visits, performed at study entry. After providing written informed consent to participate in the study, patients will be evaluated for study eligibility. The screening period includes the evaluation of inclusion criteria described above. Subjects who meet all the inclusion criteria will be enrolled.

The treatment period includes: administration of the salvage treatment PCP for 6 cycles and maintenance treatment. In order to assess the toxicity of treatment, patients will attend study centre visits at least every 2 weeks, unless clinically indicated. The response will be assessed after each cycle.

During the LTFU period, after development of confirmed PD, all patients are to be followed for survival every 1-3 months via telephone or office visit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patient with multiple myeloma who received 1 to 3 lines of treatment (including high-dose chemotherapy with stem cell support, conventional poli-chemotherapy, thalidomide- , bortezomib- and melphalan-based regimens) and is relapsed or relapsed and refractory (that means relapsed while on salvage or progression within 60 days of most recent therapy) to lenalidomide therapy.
* Patient has clinical relapse of MM based on standard criteria.
* Patient has measurable disease, defined as follows:

  * For secretory multiple myeloma, measurable disease is defined as any quantifiable serum monoclonal protein value (greater than 1 g/dL of IgG M-protein, greater than 0.5 g/dL of IgA M-protein or IgD M-protein OR urine light-chain excretion of more than 200 mg/24 hours)
  * For oligo- or non-secretory multiple myeloma, measurable disease is defined by the presence of measurable soft tissue (not bone) plasmacytomas as determined by clinical examination or applicable radiographs (i.e., MRI, CT scan).

A measurable lesion is defined as a lesion with minimum largest diameter of >20 mm (if measured by conventional techniques such as physical exam, conventional CT scan, MRI) or of >10 mm (if measured by spiral CT scan) in one dimension.

* Patient has a Karnofsky performance status ≥ 60%.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or breast feeding females.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other concomitant standard/experimental anti-myeloma drug or therapy.
* Uncontrolled or severe cardiovascular disease including myocardial infarction within 6 months of enrolment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis Other malignancy within the past 5 years. Exceptions: basal cell or non metastatic squamous cell carcinoma of the skin, cervical carcinoma in situ or FIGO Stage 1 carcinoma of the cervix.
* Concurrent medical condition or disease (e.g., active systemic infection, uncontrolled diabetes, pulmonary disease, cardiac disease) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
PCP safety and efficacy | 3 years
  We aim to identify the maximum tolerated dose (MTD) of Pomalidomide delivered in combination with Cyclophosphamide and Prednisone, defined as the dose that achieves a dose-limiting toxicity (DLT) in 25% of patients.
  The efficacy will be assessed by evaluating the very good partial response (VGPR) rate following the proposed regimen.

SECONDARY OUTCOMES:
Overall survival | 3 years
Progression-free survival | 3 years
Time-to-progression | 3 years
Time to next therapy | 3 years
Tumor response and survival in particular subgroups of patients | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza di Torino - SC Ematologia U, Torino, Italy

REFERENCES:
- [Derived] Larocca A, Montefusco V, Bringhen S, Rossi D, Crippa C, Mina R, Galli M, Marcatti M, La Verde G, Giuliani N, Magarotto V, Guglielmelli T, Rota-Scalabrini D, Omede P, Santagostino A, Baldi I, Carella AM, Boccadoro M, Corradini P, Palumbo A. Pomalidomide, cyclophosphamide, and prednisone for relapsed/refractory multiple myeloma: a multicenter phase 1/2 open-label study. Blood. 2013 Oct 17;122(16):2799-806. doi: 10.1182/blood-2013-03-488676. Epub 2013 Aug 16. PMID 23954889